CLINICAL TRIAL: NCT05942924
Title: A Randomised Trial of Repetitive Versus Selective Tactile Stimulation for Preterm Infants at Birth: The NEU-STIM Trial
Brief Title: The NEU-STIM Trial
Acronym: NEU-STIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: European Society for Paediatric Research (Unknown)
Responsible Party: Principal Investigator, Janneke Dekker, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N22.121
Record Dates: First submitted 2023-06-30; First posted 2023-07-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Infant, Premature, Diseases; Birth, Preterm
Keywords: Preterm infant; Tactile stimulation; Resuscitation
MeSH Terms: conditions — Infant, Premature, Diseases; Premature Birth

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster randomised controlled trial. The participating centre, rather than the individual infant, will be the unit of randomisation.
Who Masked: Outcomes Assessor
Masking Description: Centres will be randomised for the fortnight at which they will switch their tactile stimulation practice from selective stimulation to repetitive stimulation. The analysing researcher will be blinded for the allocation of treatment switch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective stimulation (Active Comparator): At the start of the study, selective tactile stimulation will be performed at each participating centre in accordance with international guidelines. Clinicians will gently rub the back, chest, extremities or soles of the feet if they consider the breathing of the infant to be insufficient or absent. All other procedures in the delivery room and NICU will be performed according to international and local guidelines.
  Interventions: Procedure: Selective tactile stimulation
- Repeated stimulation (Experimental): For each centre, a lot will be drawn which indicates the month in which the protocol for tactile stimulation changes from selective stimulation to repetitive stimulation.
  Repetitive stimulation is defined as gently rubbing the soles of the feet, back, chest, or extremities for 10 seconds. To prevent extinction of the stimulatory effect (reflex), every 10 second period of stimulation will be followed by 10 seconds rest (no stimulation). The repetitive stimulation will be performed for the first 5 minutes after birth, or longer if the breathing is still considered insufficient or absent. All other procedures in the delivery room and NICU will be performed according to international and local guidelines.
  Interventions: Procedure: Repeated tactile stimulation

INTERVENTIONS:
Procedure: Repeated tactile stimulation — See arm
  Arms: Repeated stimulation
Procedure: Selective tactile stimulation — See arm
  Arms: Selective stimulation

SUMMARY:
The aim of this study is to determine the effect of repetitive tactile stimulation compared to selective stimulation on oxygenation of the infant at 5 minutes after birth. Infants born before 32 weeks of gestation will be included in this trial. This is a stepped-wedge cluster randomised controlled trial. The participating centre, rather than the individual infant, will be the unit of randomisation. This design is appropriate to test the effect of an intervention that encompasses a behavioral aspect - in this case the performance of tactile stimulation.

DETAILED DESCRIPTION:
Rationale: A randomised study demonstrated that preterm infants who received repetitive stimulation at birth (10 second episodes of stroking of the soles of the feet and/or back, followed by 10 seconds rest) showed an increase in respiratory effort. This may in turn improve clinical outcomes as improved breathing effort may reduce the need for invasive respiratory support. Tactile stimulation can be immediately and easily performed at birth at no extra cost. It therefore has great potential to be implemented in delivery rooms (DRs) worldwide.

Objective: To determine the effect of repetitive tactile stimulation compared to selective stimulation on oxygenation of the infant at 5 minutes after birth.

Study design: This is a stepped-wedge cluster randomised controlled trial. The participating centre, rather than the individual infant, will be the unit of randomisation. This design is appropriate to test the effect of an intervention that encompasses a behavioral aspect - in this case the performance of tactile stimulation.

Study population: Infants born before 32 weeks of gestation will be included in this trial.

Intervention: At the start of the study, each participating centre will perform selective tactile stimulation in accordance with international guidelines, as is their usual practice. Clinicians will gently rub the back, chest, extremities or soles of the feet if they consider the breathing of the infant to be insufficient or absent. In the second stage of the study, centres will be randomised to switch their stimulation approach to repetitive stimulation. Clinicians will then gently rub the back, chest, extremities or soles of the feet for 10 seconds. To avoid extinction of the stimulatory effect (reflex), every 10 second period of stimulation will be followed by 10 seconds of rest (no stimulation). Repetitive stimulation will be performed for the first 5 minutes of life, or longer if the breathing is still considered insufficient or absent.

Main study parameter: The proportion of infants with pre-ductal oxygen saturation (SpO2) ≥ 80%.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 32 weeks of gestation can be included in this trial after parental consent.

Exclusion Criteria:

* Infants will be excluded if they are found to have a congenital abnormality or condition that has an adverse effect on breathing/ventilation or oxygenation, including: congenital diaphragmatic hernia, trachea-oesophageal fistula, cyanotic heart disease and surfactant protein deficiency. Many of the infants enrolled in the study will later be diagnosed with respiratory distress syndrome (RDS); this will not render them ineligible for inclusion.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3280 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SpO2>80 | At 5 minutes of life
  Proportion of infants with pre-ductal SpO2 >80%

SECONDARY OUTCOMES:
Heart rate | At 5 minutes after birth
  Heart rate
Number of infants who received CPAP <10min | Within 10 minutes after birth
  Number of infants who received continuous positive airway pressure
Number of infants who received PPV <10min | Within 10 minutes after birth
  Number of infants who received positive pressure ventilation
Number of infants who were intubated <10min | Within 10 minutes after birth
  Number of infants who were endotracheally intubated
Number of infants who received chest compressions <10min | Within 10 minutes after birth
  Number of infants who received chest compressions <10min
Number of infants who were administered adrenaline <10min | Within 10 minutes after birth
  Adrenaline use
Number of infants who were administered volume expansion <10min | Within 10 minutes after birth
  Number of infants who were administered volume expansion <10minv
Max FiO2 | In the first 10 minutes after birth
  Maximum FiO2
Death <10min | Within 10 minutes after birth
  Death <10min
Number of infants who were supported by CPAP in first week | In the first week after birth
  CPAP use in the NICU
Number of infants who received surfactant in first week | In the first week after birth
  Surfactant administration via INSURE, LISA or ET tube
Surfactant doses | In the first week after birth
  Number of surfactant doses administered
Number of infants who were mechanically ventilated | In the first week after birth
  Mechanical ventilation
Number of infants with abnormalities on the first cranial ultrasound | In first week after birth
  Abnormalities on first cranial ultrasound (IVH/PVL)
Death | In the first week after birth
  Mortality
Cord clamping time | During resuscitation at birth
  The time after birth at which the cord is clamped

OTHER OUTCOMES:
Congenital anomalies | At birth
  Whether the infant has congenital anomalies, e.g. diaphragmatic hernia, oesophageal atresia, cyanotic heart disease
Gestational age | At birth
  gestational age in weeks and days
Gender | At birth
  Gender of the infant
Mode of delivery | At birth
  Mode of delivery
Doses of antenatal steroids | Before birth
  Number of doses of antenatal steroids administered
Maternal magnesium sulphate | Before birth
  Whether maternal magnesium sulphate was administered
Maternal general anaesthesia | Before birth
  Whether maternal general anaesthesia was administered
Complications during pregnancy | Before birth
  Whether there were any complications during pregnancy, e.g. premature prolonged rupture of membranes, chorioamnionitis, pre-eclampsia, placental abruption, twin-to-twin transfusion syndrome, hydrops fetalis, feto-maternal haemorrhage

CONTACTS AND LOCATIONS:
Locations (43):
- Medical University of Graz, Graz, Austria
- Liège University Hospital, Liège, Belgium
- Croatia (2):
  - Clinical Hospital Center Rijeka, Rijeka
  - Clinical Center Split, Split
- Czechia (2):
  - General Faculty Hospital in Prague, Prague
  - Institute for Mother and Child Care, Prague
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Copenhagen, Copenhagen
- Germany (3):
  - University Hospital Carl Gustav Carus, Dresden
  - University Hospital Dusseldorf, Düsseldorf
  - University Hospital Tubingen, Tübingen
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Hungary (4):
  - First dept of Obstetrics and Gynaecology, Semmelweis University, Budapest
  - Second Semmelweis University, Budapest
  - University of Debrecen, Debrecen
  - Bács-Kiskun County Teaching Hospital, Szeged
- Landspitali University Hospital, Reykjavik, Iceland
- Ireland (3):
  - National Maternity Hospital, Dublin
  - Coombe Women & Infants University Hospital, Dublin
  - University Hospital Galway, Galway
- Ospedale dei Bambini Vittore Buzzi, Milan, Italy
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus MC Sophia Kinderziekenhuis, Rotterdam
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Ulleval, Oslo
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St Olav's Hospital Trondheim, Trondheim
- Poland (6):
  - Jan Biziel University Hospital No. 2 in Bydgoszcz, Bydgoszcz
  - Medical University of Gdansk, Gdansk
  - Medical University of Silesa, Katowice
  - University of Medical Sciences, Poznan
  - Provincial Hospital, Rzeszów
  - Wrocław Medical University, Wroclaw
- Hospital de Braga, Braga, Portugal
- Romania (3):
  - University Ovidius of Constanta, Constanța
  - Clinical County Emergency Hospital Sibiu, Sibiu
  - George Emil Palade University of Medicine, Târgu Mureş
- La Fe University Hospital, Valencia, Spain
- University of Health Sciences Sancaktepe Ilhan Varank Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - Bukovyna State Medical University, Chernivtsi, Chernivtsi
  - Sumy State University, Sumy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dekker J, Hooper SB, Martherus T, Cramer SJE, van Geloven N, Te Pas AB. Repetitive versus standard tactile stimulation of preterm infants at birth - A randomized controlled trial. Resuscitation. 2018 Jun;127:37-43. doi: 10.1016/j.resuscitation.2018.03.030. Epub 2018 Mar 23. PMID 29580959
- See also: Related Info — http://www.neu-stim.eu